CLINICAL TRIAL: NCT00028977
Title: A Pilot Safety, Feasibility, Efficacy And Correlative (Phase I/II) Study Assessing Herba Scutellaria Barbatae (HSB) For Metastatic Breast Cancer
Brief Title: Herbal Therapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069155; UCSF-CRO-00758; UCSF-IND-59521; NCI-G01-2043
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ban-zhi-lian; Medicine, Chinese Traditional

INTERVENTIONS:
Drug: herba scutellaria barbata
Other: herba scutellaria Barbatae (HSB)
  Other Names: Traditional Chinese Medicine

SUMMARY:
RATIONALE: The Chinese herb Scutellaria barbata contains ingredients that may slow the growth of cancer cells and may be an effective treatment for metastatic breast cancer.

PURPOSE: Phase I/II trial to study the effectiveness of Scutellaria barbata in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of Scutellaria barbata (Chinese herbal extract) in terms of tumor response in women with metastatic breast cancer.
* Determine the safety and toxicity of this therapy in these patients.
* Determine the feasibility of this therapy in these patients.
* Determine the time to progression, overall survival, and resource utilization of patients treated with this therapy.
* Determine the quality of life of patients treated with this therapy.
* Determine the bioavailability and pharmacokinetics of this therapy in these patients.

OUTLINE: Patients receive oral Scutellaria barbata (Chinese herbal extract) twice daily for 12 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer (may include original primary cancer diagnosis)
* Measurable disease
* Metastatic involvement with minimal or no symptoms

  * Solitary metastases require histological confirmation
* No extensive liver involvement (more than 50% of liver parenchyma)
* No lymphangitic pulmonary involvement
* CNS involvement or spinal cord compression allowed if stabilized by therapy for more than 3 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* More than 6 months

Hematopoietic:

* WBC at least 2,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* See Disease Characteristics
* Bilirubin no greater than 1.7 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of multiple or severe food or medicine allergies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior biologic therapy
* No concurrent anticancer biologic therapy

Chemotherapy:

* At least 1 week since prior chemotherapy
* No concurrent anticancer chemotherapy

Endocrine therapy:

* At least 1 week since prior hormonal therapy
* No concurrent anticancer hormonal therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from prior anticancer therapy
* At least 1 week since prior investigational agents
* At least 1 week since prior herbal medications
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* Concurrent pamidronate allowed
* Concurrent acupuncture or other nonherbal therapy allowed
* Concurrent nutritional vitamin supplementation (up to 5 times recommended daily allowance) allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Cancer Research Network, Incorporated, Plantation, Florida